CLINICAL TRIAL: NCT01677442
Title: Nonintubated Thoracic Epidural Anesthesia Versus Double-lumen Intubated Anesthesia in Video-assisted Thoracic Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Jun Liu, Director, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTEA001
Record Dates: First submitted 2012-05-04; First posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-04

CONDITIONS: Anaesthesia; Video Assisted Thoracic Surgery
Keywords: nonintubated; anaesthesia; VATS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no-intubated group (Experimental): Experimental: no-intubated thoracic epidural anesthesia Thoracic epidural anesthesia at the T5/T6 thoracic interspace
  Interventions: Procedure: no-intubated thoracic epidural anesthesia
- intubated group (Active Comparator): Active Comparator:double-lumen endotracheal intubated anesthesia
  Interventions: Procedure: double-lumen endotracheal intubated anesthesia

INTERVENTIONS:
Procedure: no-intubated thoracic epidural anesthesia — VATS under no-intubated thoracic epidural anesthesia
  Arms: no-intubated group
Procedure: double-lumen endotracheal intubated anesthesia — VATS under double-lumen endotracheal intubated anesthesia
  Arms: intubated group

SUMMARY:
The purpose of this study is to compare results of general Video-assisted Thoracic Surgery (VATS) operations under no-intubated thoracic epidural anesthesia (NTEA) versus those of a control group operated under general anesthesia with double-lumen endotracheal intubation.

DETAILED DESCRIPTION:
The thoracoscopic surgery always requires not only an appropriate depth of anaesthesia, but also a quiet and wide operative field. That's why anaesthesia plays a critical role in thoracoscopic surgery.

General double-lumen endotracheal intubated anesthesia with one-lung ventilation, has been accepted mandatory for Video-Assisted Thoracic Surgery (VATS) although several adverse effects can derive from this type of anesthesia like intubation-related throat injury, ventilator-induced lung injury, arrhythmia and so on. The investigators hypothesize that VATS could be performed under the no-intubated thoracic epidural anesthesia (NTEA) to avoid general anesthesia related risks.

Some cases have been reported to prove the safety and feasibility of NTEA in uncomplicated VATS. However, the comparison of NTEA and general anesthesia has been rarely investigated in such a larger magnitude number and such operation varieties. The investigators hypothesize NTEA could result in less inflammations, lower incidence of complications, less dosage of antibiotic, faster recovery eventually leading to a shorter hospital stay. For this reason, the investigators will undertaken a randomized trial comparing results of general VATS operations under NTEA versus those of a control group operated under general anesthesia with double-lumen endotracheal intubation.

A total of 500 patients will be included. The study will be performed in the first affiliated hospital of Guangzhou Medical College.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old
* signed inform consent
* Tumor size < 6 cm without right or left bronchus invasion
* Predicted FEV 1.0 > 60% or FEV1.0 > 1.5L
* EF > 50%
* PCO2 < 50mmHg,PO2 > 60mmHg（without uptaking oxygen）

Exclusion Criteria:

* Psychopath patients who cannot cooperate
* ASA score greater than 3
* A history of tuberculosis or other signs of intrapleural adhesions
* spinal malformation
* Hypovolemia or coagulation disorders
* BMI > 30
* Unfavorable reasons judged by anesthesiologist or surgeon

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
recovery time after intervention of each group | 7 days
  the time of anesthesia recovery, resumption of oral intake, and the length of hospital stay

SECONDARY OUTCOMES:
incidence of complications | 14 days

OTHER OUTCOMES:
the inflammation level | 7 days
  hemogram and some inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, Ph.D, M.D., Study Chair — Guangzhou Institute of Respiratory Disease; Jun Liu, M.D., Study Director — Guangzhou Institute of Respiratory Disease; Fei Cui, Ph.D, M.D., Principal Investigator — Guangzhou Institute of Respiratory Disease
Locations (1):
- the First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China

REFERENCES:
- See also: Related Info — http://www.gyfyy.com/